CLINICAL TRIAL: NCT02874352
Title: Incidence of Dysphagia in Intensive Care Patients With Tracheostomy Using High Resolution Pharyngoesophageal Manometry and Impedance
Brief Title: Incidence of Dysphagia in Intensive Care Patients With Tracheostomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Region Örebro County (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: JS005
Record Dates: First submitted 2016-08-17; First posted 2016-08-22 (Estimated); Last update posted 2016-08-23 (Estimated); Status verified 2016-08

CONDITIONS: Dysphagia; Oropharyngeal Dysphagia
Keywords: intensive care; tracheostomy
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- intensive care patients (Other): intensive care patients with tracheostomy/ high resolution impedance manometry with Automated Impedance Manometry analysis
  Interventions: Device: high resolution impedance manometry with Automated Impedance Manometry analysis
- healthy volunteers (Other): control group with healthy volunteers/ high resolution impedance manometry with Automated Impedance Manometry analysis
  Interventions: Device: high resolution impedance manometry with Automated Impedance Manometry analysis

INTERVENTIONS:
Device: high resolution impedance manometry with Automated Impedance Manometry analysis

SUMMARY:
This study will inform the feasibility of the High Resolution Impedance Manometry (HRIM) system combined with Automated Impedance Manometry (AIM) analysis as a screening tool for dysphagia and aspiration for the intensive care population with tracheostomy. This pilot study aims to determine the incidence of dysphagia and aspiration risk in intensive care patients with tracheostomy and the investigators hypothesise that the incidence of dysphagia in intensive care patients with tracheostomy will be higher than in an age matched population.

DETAILED DESCRIPTION:
Aspiration pneumonia is a common mechanism for recurrent mechanical ventilation episodes in intensive care patients and leads to longer hospital admissions, increased morbidity, and mortality. When length of the mechanical ventilation is prolonged the translaryngeal tube is changed to a tracheostomy tube. This practice has several advantages: further pressure damage to the vocal cords is avoided, weaning from the respirator is facilitated, and oral feeding is made possible. Swallowing difficulty, which in many cases depends on pharyngeal and upper esophageal dysfunction, is shown to be linked to aspiration pneumonia. Furthermore, previous studies indicate that swallowing dysfunction is a frequent problem in intensive care patients with tracheostomy although the reported incidence varies markedly.

Swallowing function in intensive care patients with tracheostomy is not routinely evaluated because the current diagnostic techniques, speech pathology bedside assessment (BSA), fibreoptic endoscopic evaluation of swallowing (FEES), and Videofluoroscopy (VF), are laborious, subjective expertise-dependent methods. Instead symptoms reported by the patient during fluid and food intake (cough, chest pain) are allowed to guide further feeding although it is known that silent aspiration is a common cause for aspiration pneumonia.

To prevent leakage of pharyngeal contents into the trachea most of the tracheostomy tubes are provided with an air-filled cuff. This cuff, when inflated, exerts pressure against the inner tracheal wall and thereby seals trachea around the tracheostomy tube. As security this cuff is often inflated during intake of fluids and food although there are studies that indicate this may deteriorate swallowing function and in fact increase risk for aspiration.

Automated Impedance Manometry (AIM) analysis is a method that combines measurements of manometry (pressure) and impedance (flow) using specialized equipment to generate objective numerical values indicative of the different physiological processes governing safe pharyngeal swallowing. During a swallow, these measures quantify timing of bolus flow relative to pharyngeal propulsion, any mechanical resistance to flow during propulsion, and the overall pharyngeal contractility. Pressure-flow measures are then combined to derive a swallow risk index (SRI) that provides a global assessment of swallowing and defines a level of swallowing dysfunction that may predispose to risk of aspiration. This objective assessment of swallowing function has potential to provide timely and more targeted treatment options. It is easily conducted at the bedside with minimal disruption of ongoing medical treatment, and carries with it only negligible risk to the patient. Measures are derived by using a high resolution impedance manometry (HRIM) system (Sierra Scientific Instruments, Inc., Los Angeles, California, USA). The system employs a solid state catheter with 4.2 mm outer diameter incorporating 36 circumferential 1 cm-spaced pressure sensors and 18 2-cm long impedance segments is placed transnasally with sensors straddling the entire pharyngo- and esophageal segment. Data recordings are done during several bolus swallows and analysed afterwards using AIM analysis.

Twenty intensive care patients and ten healthy volunteers are included in the study. After researchers have described the study, participants will be consented, and asked to complete a brief questionnaire about their swallow function. During the study, participants will be sitting comfortably in their bed. The manometry catheter will be passed through one nostril and down into the esophagus, stopping just at the top of the stomach. Once satisfactorily placed, the participant will be asked to swallow 4 x 5 ml; 4 x 10 ml, 3 x 20 ml of slightly salty water and 4 x 10 ml semisolid jelly. If first inflated the tracheostomy cuff is now deflated and the procedure repeated. Furthermore, part of the patients are evaluated by FEES simultaneously to HRIM measurements. Once the study is completed, the tube is removed. Patients are followed upp two months after ICU discharge with questionnaire of swallowing function and also asked to perform an additional HRIM measurement. Volunteers will perform a similar swallow series as the patients on one study occasion.

ELIGIBILITY:
Inclusion Criteria:

* Intensive care patient with tracheostomy ( applies only to patients)
* Age > 18 years
* Ability to sit upright and to swallow on command as well as to swallow thin liquids
* Informed and signed consent

Exclusion Criteria:

* Pre-existing dysphagia
* History of upper gastrointestinal surgery
* Current medication known to affect esophageal motility
* Pregnancy
* Severe coagulopathy
* Allergy to local anaesthetics

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-10; Primary Completion 2018-05 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Pressure Flow Measurements | 1 hour
  Pressure Flow measurements generated by HRIM registrations and analysed by AIM analysis

SECONDARY OUTCOMES:
Sydney Swallow Questionaire (SSQ) | 1 hour
  Clinical swallow assessment
Functional Oral Intake Scale (FOIS) | 1 hour
  Clinical swallow assessment

IPD SHARING:
Plan to Share IPD: No